CLINICAL TRIAL: NCT04276792
Title: Community Opioid Innovation Network (JCOIN): TCU Clinical Research Center
Acronym: JCOIN_TCU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Collaborators: University of New Mexico (Other); Loyola University (Other)
Responsible Party: Principal Investigator, DanicaKnight, Associate Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1UG1DA050074 (NIH)
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Addiction, Opioid
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Our design is a Hybrid Type 3 design with the primary aim to compare 2 implementation strategies, and a secondary aim to assess client-level outcomes associated with the trial; the design includes a cluster randomized parallel design with staggered starts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizontal implementation approach (Experimental): The Horizontal implementation approach of the O-TLM intervention is accompanied by facilitated collaboration between Criminal Justice and Community Behavioral Health systems. Direct involvement of stakeholders with differing perspectives and buy-in from agency leadership and policymakers are key elements. The Horizontal approach involves first developing a prototype (including how to modify existing practices, overcome implementation barriers, and manage roles and responsibilities) that are tested and refined before being rolled out systematically to other units within an agency.
  Interventions: Behavioral: TCU Opioid-Treatment Linkage Model (O-TLM)
- Vertical implementation approach (Active Comparator): The Vertical implementation approach of the O-TLM intervention relies on the traditional criminal justice system's typical use of a hierarchical structure and the use of a top-down implementation approach (i.e., administrative orders) for directing change. Top-down regulatory and policy changes are viewed as vital levers for driving system change.
  Interventions: Behavioral: TCU Opioid-Treatment Linkage Model (O-TLM)

INTERVENTIONS:
Behavioral: TCU Opioid-Treatment Linkage Model (O-TLM) — The O-TLM is focused on best practices for improving screening, identifying and linking to MOUD providers, reducing stigma, and addressing other important factors that impact justice-involved individuals returning to their communities.

SUMMARY:
There are two study periods for the TCU JCOIN project. The primary aims of Study 1 (approved by the TCU IRB) are (1) to gather information from staff on the current treatment referral process within participating communities and (2) to learn about the existing interrelationships between medical and community behavioral health (CBH) providers. TCU IRB granted approval for Phase 1 on 11/07/19, approval number: 1920-60-AM1. Study 2 (under current review by the TCU IRB) includes recruitment across 18 community collaboration sites across 3 states; these communities will participate in the TCU Opioid-Treatment Linkage Model (O-TLM) protocol. The O-TLM is focused on best practices for improving screening, identifying and linking to MOUD providers, reducing stigma, and addressing other important factors that impact justice-involved individuals returning to their communities. Along with their agency records, information collected from justice-involved individuals within the target communities will be examined to assess O-TLM impact on improving public health and public safety outcomes. Furthermore, stakeholder staff across community organizations, including criminal justice and treatment agencies, will be asked to complete surveys on the O-TLM regarding its acceptability and adoption, as well as on best training strategies.

ELIGIBILITY:
Inclusion Criteria:

* client level participant eligibility includes having a history of opioid use or at risk for opioid use; being released to a participating community while under supervision
* staff level participant eligibility includes being a key member of a participating community and involved in the service assessment and referral process of justice-involved individuals.

Exclusion Criteria:

* no history of opioid use or being at risk of opioid use; not being released to a participating community.
* staff level participant exclusion criteria include not being a key member of a participating community and not being involved in the service assessment and referral process of justice-involved individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Public Health assessed by decrease in days and amount of illicit drug use, including opioids | 6 months and 12 months post-release
  decreases in days and amount of illicit drug use, including opioids assessed through client interviews using the timeline follow-back method
Public Safety as assessed through reduction in rearrest rates | 6 months and 12 months post-release
  reductions in rearrest rates measured through justice and department of pubic safety records
Increase in Access to Services | 6 months and 12 months post-release
  referral rate increase as self-reported through client interviews and provided through justice records
Increase in Retention in Services | 6 months and 12 months post-release
  appointments kept as self-reported through client interviews and provided through justice and provider records

SECONDARY OUTCOMES:
Systems Impact as assessed through improved intervention attitudes | 6 and 12 months post implementation start
  staff attitudes of intervention acceptability as assessed through survey
Systems Impact as assessed through intervention cost | 6 and 12 months post implementation start
  accumulated cost of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Danica K Knight, PhD, Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Will adhere to NIH JCOIN approved plan
Supporting Information: Study Protocol, ICF